CLINICAL TRIAL: NCT04616521
Title: Asymmetric Deep Brain Stimulation for Parkinson's Disease: A Multicenter, Prospective, Single Arm, Open Label Study
Brief Title: Asymmetric DBS for PD : A Multicenter, Prospective, Single Arm, Open Label Study
Acronym: ADP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Huashan Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); West China Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Tianjin Huanhu Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of Center for Functional Neurosurgery, Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ruijin_ADP
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Parkinson Disease
Keywords: deep brain stimulation; subthalamic nucleus; globus pallidus interna; asymmetric deep brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Asymmetric DBS group (Experimental): In this arm, a one-staged combined unilateral STN and contralateral GPi DBS will be implanted into PD patients. For postural instability and gait difficulty (PIGD)-dominant patients, the GPi in the side contralateral to the leg with longer step length will be targeted. For tremor-dominant (TD) patients, the STN in the side contralateral to the body side that mostly affected will be targeted. For PD patients of mixed type, the choice of target will depend on the judgement of a multidisciplinary team based on clinical features.
  Interventions: Procedure: Deep brain stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation — The surgical intervention named deep brain stimulation is a well-established neurosurgical treatment for moderate-to-advanced stage PD. The targets used in this study are STN and GPi, which are widely accepted and used for symptom control in PD. The devices used for intervention have been approved by Chinese National Medical Products Administration (CFDA). The postoperative drug dosage adjustment depends on the efficacy of DBS and the judgment of the movement disorder specialist.

SUMMARY:
Deep brain stimulation (DBS) is an efficacious neurosurgical treatment for moderate-to-late stage Parkinson's disease (PD). The subthalamic nucleus (STN) and globus pallidus interna (GPi) are two targets extensively studied and used worldwide in treating PD. Although the conventional SYMMETRIC bilateral STN and GPi DBS are shown to be effective in controlling motor symptoms such as bradykinesia, tremor, and dyskinesia, each target has its pros and cons in terms of axial symptom control, medication reduction, cognitive decline, and programming. Therefore, we speculate that an ASYMMETRIC bilateral implantation of DBS leads (i.e., combined unilateral STN and contralateral GPi DBS) may be able to bring the greatest clinical benefits to PD patients by taking advantage of both bilateral STN and GPi DBS at the same time. The preliminary retrospective study containing eight PD patients undergoing asymmetric implantation of DBS demonstrated the safety and efficacy of this treatment strategy during short-term follow-up. This multicenter, single arm, open label study aims to prospectively investigate during the long-term follow-up the safety and efficacy of asymmetric DBS for PD in terms of motor and nonmotor symptoms, medication reduction, cognitive decline, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease based on the MDS clinical diagnostic criteria for Parkinson's disease
* Aged more than 18 years
* Levodopa challenge test indicating a preoperative levodopa responsiveness over 24% based on MDS UPDRS-III
* the modified Hoehn-Yahr Scale between 2 and 4 under on-medication condition
* Compliance with written informed consent

Exclusion Criteria:

* Atypical parkinsonian syndrome
* History of stroke, encephalitis, neuroleptic uses, MRI scan with evidence of significant brain atrophy, lacunar infracts, or other conditions that might interfere with the intracranial surgery
* Presence of cognitive, or psychiatric or other co-morbidities (e.g., dementia, epilepsy, cranial traumatism, brain tumor, schizophrenia, severe depression or bipolar disorder, personality disorder, etc.) that might interfere with the patient's ability to complete the evaluations or to provide informed consent
* Presence of anatomical abnormalities in the target region
* Clinically significant medical history or that increases pre-/post-operative complications
* Other conditions considered by the investigators that might interfere with the surgery procedure, the follow-ups, and the interpretation of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale - Part III (MDS UPDRS-III) | Followed for minimum of 7 years
  Score ranges from 0 to 132, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale - Part I, II, IV | Followed for minimum of 7 years
  Score ranges from 0 to 128, higher scores mean a worse outcome.
Time-Up-Go (TUG) task | Followed for minimum of 7 years
Berg Balance Scale, BBS | Followed for minimum of 7 years
  Score ranges from 0 to 132, higher scores mean a better outcome.
Gait and Falls Questionnaire, GFQ | Followed for minimum of 7 years
  Score ranges from 0 to 64, higher scores mean a worse outcome.
Montreal Cognitive Assessment (MoCA) | Followed for minimum of 7 years
Beck Depression Inventory, BDI | Followed for minimum of 7 years
Beck Anxiety Inventory, BAI | Followed for minimum of 7 years
Apathy Estimation Scale, AES | Followed for minimum of 7 years
Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Current Full, QUIP-CF | Followed for minimum of 7 years
  True-or-false questions screening the obsessive-compulsive behaviors in parkinson's disease
Epworth Sleepiness Scale, ESS | Followed for minimum of 7 years
Non-Motor Symptoms Scale, NMSS | Followed for minimum of 7 years
  Score ranges from 0 to 360, higher scores mean a worseoutcome.
Scales for Outcomes in PArkinson's disease - Autonomic, SCOPA-AUT | Followed for minimum of 7 years
8-item Parkinson's Disease Questionnaire (PDQ-8) | Followed for minimum of 7 years
5-Level EuroQol Five Dimensions Questionnaire, EQ-5D-5L | Followed for minimum of 7 years
Levodopa Equivalent Daily Dose, LEDD | Followed for minimum of 7 years
Adverse Events, Severe Adverse Events | Followed for minimum of 7 years